CLINICAL TRIAL: NCT01043185
Title: A Double-blind, Placebo Controlled, Randomised, Phase IIA Pharmacodynamic 4-way Cross-over Study to Estimate the Dose Response Relationship of AZD3355 on the Number of Reflux Episodes Assessed by Impedance/pH in Patients With GERD and a Partial Response to PPI Treatment
Brief Title: A Study to Estimate Effect of 4 Different Doses of AZD3355 on Reflux Episodes, Which Patients With Gastroesophageal Reflux Disease (GERD) May Experience
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D9120C00032
Record Dates: First submitted 2009-12-22; First posted 2010-01-06 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; lesogaberan; impedance; pH; pharmacokinetics; safety; tolerability
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — lesogaberan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): AZD3355 30 mg
  Interventions: Drug: AZD3355
- B (Experimental): AZD3355 90 mg
  Interventions: Drug: AZD3355
- C (Experimental): AZD3355 120 mg
  Interventions: Drug: AZD3355
- D (Experimental): AZD3355 240 mg
  Interventions: Drug: AZD3355
- E (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AZD3355 — 30 mg orally in the morning and 30 mg in the evening for 1 day
  Arms: A
Drug: AZD3355 — 90 mg orally in the morning and 90 mg in the evening for 1 day
  Arms: B
Drug: AZD3355 — 120 mg orally in the morning and 120 mg in the evening for 1 day
  Arms: C
Drug: AZD3355 — 240 mg orally in the morning and 240 mg in the evening for 1 day
  Arms: D
Drug: placebo — Placebo capsules orally in the morning and placebo capsules in the evening for 1 day
  Arms: E

SUMMARY:
The purpose of the study is to estimate what effect 4 different doses of AZD3355 will have on the number of reflux episodes, in patients who have GERD and still experience symptoms despite proton pump inhibitor (PPI) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* History of GERD with persistent symptoms despite treatment with PPI
* Otherwise normal physical health

Exclusion Criteria:

* History of GERD with symptoms that has not improved at all during treatment with PPI
* Prior surgery of the upper gastrointestinal tract
* History of significant heart disease, cardiovascular, respiratory, hepatic, renal, metabolic, psychiatric or gastrointestinal disorders besides GERD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Miner, Principal Investigator — Oklahoma Foundation of Digestive Research; Debra G Silberg, Study Director — AstraZeneca
Locations (1):
- Research Site, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Miner PB Jr, Silberg DG, Ruth M, Miller F, Pandolfino J. Dose-dependent effects of lesogaberan on reflux measures in patients with refractory gastroesophageal reflux disease: a randomized, placebo-controlled study. BMC Gastroenterol. 2014 Nov 18;14:188. doi: 10.1186/1471-230X-14-188. PMID 25407279

RESULTS

PARTICIPANT FLOW:
Groups:
- First 30mg, Then 90mg, Then 120mg, Then Placebo: Period 1: AZD3355 30mg. Period 2: AZD3355 90mg. Period 3: AZD3355 120mg. Period 4: placebo. Morning and evening dose in each period.
- First 30mg, Then 90mg, Then Placebo, Then 120mg: Period 1: AZD3355 30mg. Period 2: AZD3355 90mg. Period 3: placebo. Period 4: AZD3355 120mg. Morning and evening dose in each period.
- First 120mg, Then Placebo, Then 240mg, Then 90mg: Period 1: AZD3355 120mg. Period 2: placebo. Period 3: AZD3355 240mg. Period 4: AZD3355 90mg. Morning and evening dose in each period.
- First Placebo, Then 30mg, Then 90mg, Then 120mg: Period 1: placebo. Period 2: AZD3355 30mg. Period 3: AZD3355 90mg. Period 4: AZD3355 120mg. Morning and evening dose in each period.
- First 90mg, Then Placebo, Then 120mg, Then 240mg: Period 1: AZD3355 90mg. Period 2: placebo. Period 3: AZD3355 120mg. Period 4: AZD3355 240mg. Morning and evening dose in each period.
- First Placebo, Then 240mg, Then 90mg, Then 30mg: Period 1: placebo. Period 2: AZD3355 240mg. Period 3: AZD3355 90mg. Period 4: AZD3355 30mg. Morning and evening dose in each period.
- First 90mg, Then 120mg, Then Placebo, Then 240mg: Period 1: AZD3355 90mg. Period 2: AZD3355 120mg. Period 3: placebo. Period 4: AZD3355 240mg. Morning and evening dose in each period.
- First 120mg, Then 30mg, Then 240mg, Then Placebo: Period 1: AZD3355 120mg. Period 2: AZD3355 30mg. Period 3: AZD3355 240mg. Period 4: placebo. Morning and evening dose in each period.
- First 240mg, Then 30mg, Then 90mg, Then Placebo: Period 1: AZD3355 240mg. Period 2: AZD3355 30mg. Period 3: AZD3355 90mg. Period 4: placebo. Morning and evening dose in each period.
- First Placebo, Then 120mg, Then 30mg, Then 240mg: Period 1: placebo. Period 2: AZD3355 120mg. Period 3: AZD3355 30mg. Period 4: AZD3355 240mg. Morning and evening dose in each period.
Period: Period 1 - First Intervention
Arm/Group | First 30mg, Then 90mg, Then 120mg, Then Placebo | First 30mg, Then 90mg, Then Placebo, Then 120mg | First 120mg, Then Placebo, Then 240mg, Then 90mg | First Placebo, Then 30mg, Then 90mg, Then 120mg | First 90mg, Then Placebo, Then 120mg, Then 240mg | First Placebo, Then 240mg, Then 90mg, Then 30mg | First 90mg, Then 120mg, Then Placebo, Then 240mg | First 120mg, Then 30mg, Then 240mg, Then Placebo | First 240mg, Then 30mg, Then 90mg, Then Placebo | First Placebo, Then 120mg, Then 30mg, Then 240mg
Started | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 - First Washout Period
Arm/Group | First 30mg, Then 90mg, Then 120mg, Then Placebo | First 30mg, Then 90mg, Then Placebo, Then 120mg | First 120mg, Then Placebo, Then 240mg, Then 90mg | First Placebo, Then 30mg, Then 90mg, Then 120mg | First 90mg, Then Placebo, Then 120mg, Then 240mg | First Placebo, Then 240mg, Then 90mg, Then 30mg | First 90mg, Then 120mg, Then Placebo, Then 240mg | First 120mg, Then 30mg, Then 240mg, Then Placebo | First 240mg, Then 30mg, Then 90mg, Then Placebo | First Placebo, Then 120mg, Then 30mg, Then 240mg
Started | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 - Second Intervention
Arm/Group | First 30mg, Then 90mg, Then 120mg, Then Placebo | First 30mg, Then 90mg, Then Placebo, Then 120mg | First 120mg, Then Placebo, Then 240mg, Then 90mg | First Placebo, Then 30mg, Then 90mg, Then 120mg | First 90mg, Then Placebo, Then 120mg, Then 240mg | First Placebo, Then 240mg, Then 90mg, Then 30mg | First 90mg, Then 120mg, Then Placebo, Then 240mg | First 120mg, Then 30mg, Then 240mg, Then Placebo | First 240mg, Then 30mg, Then 90mg, Then Placebo | First Placebo, Then 120mg, Then 30mg, Then 240mg
Started | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 - Second Washout Period
Arm/Group | First 30mg, Then 90mg, Then 120mg, Then Placebo | First 30mg, Then 90mg, Then Placebo, Then 120mg | First 120mg, Then Placebo, Then 240mg, Then 90mg | First Placebo, Then 30mg, Then 90mg, Then 120mg | First 90mg, Then Placebo, Then 120mg, Then 240mg | First Placebo, Then 240mg, Then 90mg, Then 30mg | First 90mg, Then 120mg, Then Placebo, Then 240mg | First 120mg, Then 30mg, Then 240mg, Then Placebo | First 240mg, Then 30mg, Then 90mg, Then Placebo | First Placebo, Then 120mg, Then 30mg, Then 240mg
Started | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5 - Third Intervention
Arm/Group | First 30mg, Then 90mg, Then 120mg, Then Placebo | First 30mg, Then 90mg, Then Placebo, Then 120mg | First 120mg, Then Placebo, Then 240mg, Then 90mg | First Placebo, Then 30mg, Then 90mg, Then 120mg | First 90mg, Then Placebo, Then 120mg, Then 240mg | First Placebo, Then 240mg, Then 90mg, Then 30mg | First 90mg, Then 120mg, Then Placebo, Then 240mg | First 120mg, Then 30mg, Then 240mg, Then Placebo | First 240mg, Then 30mg, Then 90mg, Then Placebo | First Placebo, Then 120mg, Then 30mg, Then 240mg
Started | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 6 - Third Washout Period
Arm/Group | First 30mg, Then 90mg, Then 120mg, Then Placebo | First 30mg, Then 90mg, Then Placebo, Then 120mg | First 120mg, Then Placebo, Then 240mg, Then 90mg | First Placebo, Then 30mg, Then 90mg, Then 120mg | First 90mg, Then Placebo, Then 120mg, Then 240mg | First Placebo, Then 240mg, Then 90mg, Then 30mg | First 90mg, Then 120mg, Then Placebo, Then 240mg | First 120mg, Then 30mg, Then 240mg, Then Placebo | First 240mg, Then 30mg, Then 90mg, Then Placebo | First Placebo, Then 120mg, Then 30mg, Then 240mg
Started | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 7 - Fourth Intervention
Arm/Group | First 30mg, Then 90mg, Then 120mg, Then Placebo | First 30mg, Then 90mg, Then Placebo, Then 120mg | First 120mg, Then Placebo, Then 240mg, Then 90mg | First Placebo, Then 30mg, Then 90mg, Then 120mg | First 90mg, Then Placebo, Then 120mg, Then 240mg | First Placebo, Then 240mg, Then 90mg, Then 30mg | First 90mg, Then 120mg, Then Placebo, Then 240mg | First 120mg, Then 30mg, Then 240mg, Then Placebo | First 240mg, Then 30mg, Then 90mg, Then Placebo | First Placebo, Then 120mg, Then 30mg, Then 240mg
Started | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 3
Completed | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all groups randomized to one of 10 sequences of drug or placebo.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 27
Age Continuous [Mean (Full Range); unit: Years] | 43.3 [18 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Reflux Episodes During 24 Hours
Description: Number of reflux episodes assessed during ambulatory impedance-pH recording (defined as starting with a drop in impedance to below 50% of baseline and ending when impedance recovers to above 50% of baseline)
Time Frame: Measured during 24 hours at 4 different visits with a 7-28 days interval between
Population: Efficacy Analysis Set (EAS). From the safety analysis set with 27 patients, the EAS excludes 2 patients; 1 due to a positive drug of abuse screen and 1 due to poor quality of the impedance/pH tracings during all 4 study periods. Additionally, 3 patients were partly excluded from the EAS due to poor quality of the tracings during 1 study period.
Measure: Geometric Mean (95% Confidence Interval); unit: Episodes
Groups:
- AZD3355 30 mg: a morning and an evening dose of AZD3355 30 mg
- AZD3355 90 mg: a morning and an evening dose of AZD3355 90 mg
- AZD3355 120 mg: a morning and an evening dose of AZD3355 120 mg
- AZD3355 240 mg: a morning and an evening dose of AZD3355 240 mg
- Placebo: a morning and an evening dose of placebo
Arm/Group | AZD3355 30 mg | AZD3355 90 mg | AZD3355 120 mg | AZD3355 240 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 20 | 18 | 24
Episodes | 59.4 [49.1 to 71.8] | 50.7 [41.8 to 61.4] | 44.3 [36.9 to 53.2] | 38.0 [31.4 to 46.0] | 80.5 [67.5 to 96.1]

2. Secondary Outcome: Number of Acid Reflux Episodes
Description: Number of reflux episodes as defined for the primary outcome measure with an intraesophageal pH <4 (or a drop of at least 1 pH unit if pH is already <4) lasting more than 5 s.
Time Frame: Measured during 24 hours at 4 different visits with a 7-28 days interval between
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Episodes
Arm/Group | AZD3355 30 mg | AZD3355 90 mg | AZD3355 120 mg | AZD3355 240 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 20 | 18 | 24
Episodes | 9.6 [4.9 to 18.8] | 8.0 [4.1 to 15.8] | 6.2 [3.2 to 12.0] | 6.3 [3.2 to 12.4] | 14.7 [7.7 to 28.0]

3. Secondary Outcome: Number of Weakly Acidic Reflux Episodes
Description: Number of reflux episodes as defined for the primary outcome measure with an intraesophageal pH 4.0-6.5 lasting more than 5 s.
Time Frame: Measured during 24 hours at 4 different visits with a 7-28 days interval between
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Episodes
Arm/Group | AZD3355 30 mg | AZD3355 90 mg | AZD3355 120 mg | AZD3355 240 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 20 | 18 | 24
Episodes | 37.0 [27.4 to 49.9] | 35.4 [26.2 to 47.8] | 28.7 [21.5 to 38.3] | 28.4 [21.0 to 38.3] | 51.6 [39.0 to 68.2]

4. Secondary Outcome: Number of Weakly Alkaline Reflux Episodes
Description: Number of reflux episodes as defined for the primary outcome measure with an intraesophageal pH ≥6.5 lasting more than 5 s.
Time Frame: Measured during 24 hours at 4 different visits with a 7-28 days interval between
Population: as for outcome 1
Measure: Median (Full Range); unit: Episodes
Arm/Group | AZD3355 30 mg | AZD3355 90 mg | AZD3355 120 mg | AZD3355 240 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 20 | 18 | 24
Episodes | 0 [0 to 0] | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 2] | 0 [0 to 1]

ADVERSE EVENTS:
Arm/Group | AZD3355 30 mg | AZD3355 90 mg | AZD3355 120 mg | AZD3355 240 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/21 | 1/20 | 0/26
Other Adverse Events (participants affected / at risk) | 0/19 | 1/21 | 0/21 | 3/20 | 2/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD3355 30 mg (N=19) | AZD3355 90 mg (N=21) | AZD3355 120 mg (N=21) | AZD3355 240 mg (N=20) | Placebo (N=26)
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD3355 30 mg (N=19) | AZD3355 90 mg (N=21) | AZD3355 120 mg (N=21) | AZD3355 240 mg (N=20) | Placebo (N=26)
Gastroenteritisviral (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between PI and Sponsor (AZ) or its agents that restricts the PI's right to discuss/publish trial results after the trial is completed.The PI agrees to collaborate in good faith with AZ with regards to content and formation of any publication or disclosure to be made by PI and to pay due consideration to opinions offered by AZ.